CLINICAL TRIAL: NCT05564000
Title: A Study of Bystander Intention and Behavior to Prevent Dating Violence Among College Students --Application of the Theory of Planned Behavior to Explore, Construct and Evaluate Dating Violence Education Programs (Second to the Third Year)
Brief Title: Effects of Dating Violence Education Program on Bystanders' Help-giving Intention and Behavior Among College Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20200054; MOST 110-2410-H-037-005-SS2 (Other Grant/Funding Number: MOST)
Record Dates: First submitted 2022-09-20; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Intimate Partner Violence
Keywords: dating violence; bystander education program; attitude; self-efficacy; intention; behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: experimental and control group
Who Masked: Outcomes Assessor
Masking Description: The principal investigator (outcomes assessor) does not know who participate in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: accept three weeks Dating Violence Prevention Program online; every week 20-30 minutes.
  The measurements of dating violence myths, bystander attitude, subjective norm, self-efficacy, intention, and behavior were implemented with a pre-, post-test, and 2-month follow-up design to analyze the immediate and continued educational effects.
  Interventions: Other: Dating Violence Prevention Program
- Control group (No Intervention): Control group: no intervention. The measurements of dating violence myths, bystander attitude, subjective norm, self-efficacy, intention, and behavior were implemented with a pre-, post-test, and 2-month follow-up.

INTERVENTIONS:
Other: Dating Violence Prevention Program — We designed and constructed the e-learning platform as an education program on dating violence based on the theory of planned behavior to evaluate the effectiveness of the programs in improving dating violence myths, bystander help-giving attitude, subjective norms, self-efficacy, intention, and behavior.
  Arms: Experimental group

SUMMARY:
The present study was a quasi-experiment study. College students were recruited and divided into two groups: the experimental group and the control group. There were roughly 180-210 participants in each group, which totaled 360-420 people in all. The measurements of Dating Violence Myths and Dating Violence Bystander Help-giving Intention Questionnaire were implemented with a pre-, post-test, and 2-month follow-up design to analyze the immediate and continued educational effects. The investigators also invite 10 -30 participants to participate in online anonymous group interviews to collect qualitative data. The investigators expect dating violence education programs can improve college students' dating violence myths and dating violence bystander help-giving intention and behavior. The dating violence education program on the e-learning platform can be widely used in other colleges to build up safe dating relationships and friendly campuses.

DETAILED DESCRIPTION:
Dating violence is a global health problem that strongly affects young people's physical and mental health. Whether bystanders who are witnesses or are asked for help take action to help victims influences the cycle of violence, but the studies of bystander behavior and prevention programs for dating violence have lacked in Taiwan. The investigators designed and constructed the e-learning platform as an education program on dating violence based on the theory of planned behavior to evaluate the effectiveness of the programs in improving dating violence myths and bystanders' help-giving intention and behavior among college students. The present study was a quasi-experiment study. College students were recruited and divided into two groups: the experimental group and the control group. There were roughly 180-210 participants in each group, which totaled 360-420 people in all. The measurements of Dating Violence Myths and Dating Violence Bystander Help-giving Intention Questionnaire were implemented with a pre-, post-test, and 2-month follow-up design to analyze the immediate and continued educational effects. The investigators also invite 10 -30 participants to participate in online anonymous group interviews to collect qualitative data. The investigators expect dating violence education programs can improve college students' dating violence myths and dating violence bystander help-giving intention and behavior. The dating violence education program on the e-learning platform can be widely used in other colleges to build up safe dating relationships and friendly campuses.

ELIGIBILITY:
Inclusion Criteria:

* College students aged 18-25 years, and agree to participate in this study.

Exclusion Criteria:

* Married college students.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Dating Violence Myths Scale | at first week before dating violence education program
  Dating Violence Myths Scale will be used to evaluate the individual level of inaccurate or or false beliefs about dating violence (including physical, mental, and sexual violence) in experimental and control group.
Dating Violence Myths Scale | at second week after dating violence education program
  Dating Violence Myths Scale will be used to evaluate the individual level of inaccurate or false beliefs about dating violence (including physical, mental, and sexual violence) in experimental and control group.
Dating Violence Myths Scale | at two months after dating violence education program
  Dating Violence Myths Scale will be used to evaluate the individual level of inaccurate or false beliefs about dating violence (including physical, mental, and sexual violence) in experimental and control group.
Dating Violence Bystander Help-giving Intention Questionnaire (DVBHIQ) | at first week before dating violence education program
  DVBHIQ will be used to assess the individual help-giving intention toward victims suffering dating violence in experimental and control group.
Dating Violence Bystander Help-giving Intention Questionnaire | at second week after dating violence education program
  DVBHIQ will be used to assess the individual help-giving intention toward victims suffering dating violence in experimental and control group.
Dating Violence Bystander Help-giving Intention Questionnaire | at two months after dating violence education program
  DVBHIQ will be used to assess the individual help-giving intention toward victims suffering dating violence in experimental and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Li Hou, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No